CLINICAL TRIAL: NCT07208201
Title: Clinical Utility of Bronchoalveolar Lavage in Interstitial Lung Diseases
Brief Title: Bronchoalveolar Lavage in Interstitial Lung Diseases to Characterization of Specific Inflammatory Cellular Infiltrate in Different Interstitial Lung Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Maha Ahmed Abd EL Gawad Mohammed Okasha (Other)
Responsible Party: Sponsor-Investigator, Maha Ahmed Abd EL Gawad Mohammed Okasha, pulmonologist at Assiut Police hospital, Assiut University
Organization: Assiut University (Other)
Other Study IDs: BAL in ILD
Record Dates: First submitted 2025-09-01; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Interstitial Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bronchoscopy — BAL is performed with the fiberoptic bronchoscope in a wedge position within the selected bronchopulmonary segment.
  The total instilled volume of normal saline should be no less than 100 ml and should not exceed 300 ml.
  Three to five sequentially instilled aliquots are generally withdrawn after each aliquot instillation.
  For optimal sampling of distal airspaces, the total volume (pooled aliquots) retrieved should be greater than or equal to 30% of the total instilled volume.
  A total volume of retrieved fluid less than 30% may provide a misleading cell differential, especially if total retrieved volume is less than 10% of total instilled volume.
  If less than 5% of each instilled aliquot volume is recovered during the procedure due to retention of most of the fluid in the lavaged segment, the procedure should be aborted to avoid increased risk of tissue disruption and/or inflammatory mediator release due to overdistention of the lavaged segment.

SUMMARY:
Interstitial lung disease (ILD) represents a various group of disorders characterized by inflammation and fibrosis within the lung parenchyma.[1] ILD refers to a group of diffuse parenchymal lung disorders, including a spectrum of conditions such as idiopathic pulmonary fibrosis (IPF), sarcoidosis, and connective tissue disease-associated ILD (CTD-ILD) characterized by inflammation and fibrosis of the interstitium.

ILD results in Impaired lung function and, in severe cases, respiratory failure.[1] Diagnosing ILD is a complex task due to the heterogeneous nature of these disorders.

Distinguishing between different ILD subtypes and identifying disease progression present ongoing challenges in clinical practice. .[2] BAL emerges as a key investigative tool , allowing for the collection of bronchoalveolar fluid.

The cellular and molecular composition of BAL fluid provides valuable insights into the underlying pathology, aiding in the differential diagnosis of ILD subtypes.

The gold standard in BAL analysis is cytological examination by microscopy.[3] Flow cytometry is an updated method of BAL analysis which can provide quicker and more objective results and, with the appropriate design of antibody panels, accurately quantify the main leukocyte subsets.

Several studies have described the usefulness of flowcytometry for the discrimination of sarcoidosis from other lymphocytic pathologies or even to perform leukocyte subset counting in diverse ILDs.[4][5]

Both microscopic and flowcytometric examination of BAL in ILD are complementary tools that provide comprehensive information about the cellular landscape of the lower respiratory tract ,conclusive for:

Accurate diagnosis

Primary aim:

Characterization of specific inflammatory cellular infiltrate in different interstitial lung diseases.

- Secondary aims:

1. Correlation between clinical ,radiological and inflammatory cellular pattern as regards BAL findings of different interstitial lung diseases
2. Assessment of impact on outcome, prognosis and survival of the disease as regards management modification after BAL characterization

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical suspicion of ILD based on symptoms, clinical examination, and radiological findings or newly diagnosed cases .
* HRCT findings consistent with ILD
* Willingness to undergo bronchoscopy with BAL and provide informed consent

Exclusion Criteria:

* Hemodynamic instability or ICU admission at time of evaluation
* Oxygen saturation < 88% on room air or < 92% on oxygen therapy
* Absolute contraindications to bronchoscopy (e.g., uncorrected bleeding diathesis, recent myocardial infarction)
* Associated chronic chest diseases other than ILD (COPD. bronchial asthma and lung cancer )
* Known active pulmonary infection or recent antibiotic treatment (< 2 weeks)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subtypes of interstitial lung diseases
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-12-04 (Estimated); Primary Completion 2026-12-04 (Estimated); Study Completion 2027-12-04 (Estimated)

PRIMARY OUTCOMES:
description of pattern and percentage of specific inflammatory cellular infiltrate in different interstitial lung diseases in bronchoalveolar lavage . | 2 years